CLINICAL TRIAL: NCT00445952
Title: Fungemia Survey in Cancer Patients
Brief Title: Natural History Study of Fungal Infections of the Blood in Patients With Cancer or in Patients Who Have Undergone a Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-65031; EORTC-65031
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cancer
Keywords: breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; male breast cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; unspecified adult solid tumor, protocol specific; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; contiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I small lymphocytic lymphoma; stage I marginal zone lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; refractory multiple myeloma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; relapsing chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; acute undifferentiated leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; refractory hairy cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; post-transplant lymphoproliferative disorder; extramedullary plasmacytoma; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult grade III lymphomatoid granulomatosis; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; meningeal chronic myelogenous leukemia; primary central nervous system non-Hodgkin lymphoma; stage I adult Hodgkin lymphoma; adult nasal type extranodal NK/T-cell lymphoma; infection; limited stage small cell lung cancer; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Neoplasms; Breast Carcinoma In Situ; Breast Neoplasms; Breast Neoplasms, Male; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Congenital Abnormalities; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Multiple Myeloma; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Waldenstrom Macroglobulinemia; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Lymphoma, Extranodal NK-T-Cell; Infections; Leukemia, Large Granular Lymphocytic | interventions — Watchful Waiting

INTERVENTIONS:
Other: clinical observation
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Gathering information about how often fungal infections of the blood occur in patients with cancer or in patients who have undergone stem cell transplant may help doctors learn more about the disease.

PURPOSE: This natural history study is collecting information about fungal infections of the blood over time from patients with cancer or from patients who have undergone a stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of fungemia in relation to the number of admissions to the hospital in patients with solid tumor or hematologic malignancy or in patients who have undergone hematopoietic stem cell transplantation.
* Determine the fungal species distribution, prognostic factors for outcome, and crude and attributable mortality in patients also diagnosed with fungemia.

OUTLINE: This is a multicenter, nonrandomized, prospective study.

* Group A (no documented fungemia at study entry): Data regarding the number of patients with cancer or who have undergone hematopoietic stem cell transplantation, including those who develop documented fungemia, who are admitted to the hospital is collected for 2 years.
* Group B (documented fungemia at study entry): Fungal strains isolated from the initial positive blood culture are collected and undergo examination, including confirmation of species identification, susceptibility testing, and/or minimum inhibitory concentration determination. Data, including antifungal treatment, clinical and microbiological response to antifungal treatment (at 2, 4, and 12 weeks after diagnosis), and survival status, is collected for each documented fungemia episode* for up to 12 weeks after diagnosis of fungemia.

NOTE: *That occurs within a 2-year period.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Group A:

  * Meets any of the following criteria:

    * Diagnosis of hematological malignancy including, but not limited to, any of the following:

      * Acute lymphoblastic leukemia
      * Acute myeloid leukemia
      * Myelodysplastic syndromes
      * Chronic lymphocytic leukemia
    * Diagnosis of solid tumor, including, but not limited to, any of the following:

      * Breast cancer (hormone receptor status not specified)
      * Lung cancer
      * Colon cancer
    * Recipient of a hematopoietic stem cell transplantation, including, but not limited to, any of the following:

      * Allogeneic or autologous bone marrow transplantation
      * Peripheral blood stem cell transplantation
  * Admitted to a participating hospital ward (defined as ≥ 1 overnight stay)
* Group B:

  * Meets the same criteria as in group A
  * Positive blood culture for a fungus

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior participation in this study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
Relative incidence of fungemia
Fungal species distribution
Survival in patients with fungemia
Mortality at 2, 4, and 12 weeks after diagnosis of fungemia

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, Study Chair — German Hodgkin's Lymphoma Study Group
Locations (5):
- Institut Jules Bordet, Brussels, Belgium
- CHU de Grenoble - Hopital de la Tronche, Grenoble, France
- German Hodgkin's Lymphoma Study Group, Cologne, Germany
- Ospedale San Martino, Genoa, Italy
- Hopital Cantonal Universitaire de Geneve, Geneva, Switzerland